CLINICAL TRIAL: NCT06267989
Title: The Effectiveness and Cost-effectiveness of Early Intervention to Correct the Position of a Palatally Displaced Maxillary Permanent Canine: A Multicentre RCT
Brief Title: The Effectiveness of Early Intervention to Correct the Position of PDC:s
Acronym: PDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Sheffield (Other); Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gothenburg University/Göteborg
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Ectopic Tooth Eruption; Palatal Expansion Technique; Randomized Clinical Trial
MeSH Terms: conditions — Tooth Eruption, Ectopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extraction (Active Comparator): Extraction of the primary canine
  Interventions: Procedure: Extraction of the primary canine teeth
- Expansion (Experimental): Rapid maxillary expansion without extraction of the primary canine
  Interventions: Procedure: Expansion
- Control (No Intervention): No intervention during the observation period (18 months)

INTERVENTIONS:
Procedure: Extraction of the primary canine teeth — Extraction of the primary teeth has show to be successful in some cases.
  Other Names: Extraction of the baby teeth
  Arms: Extraction
Procedure: Expansion — Expansion of the maxilla with rapid maxillary expander with no extractions
  Arms: Expansion

SUMMARY:
Approximately 2-3% of children will have problems with one or both of their permanent or 'adult' canine teeth in the upper jaw. These canine teeth sometimes fail to erupt properly, because they are displaced into the roof of the mouth or palate. These are known as palatally displaced canines, PDC, (Brin et al., 1986, Ericson and Kurol, 1987). In addition to failing to erupt, displaced teeth can cause problems, such as damage to the roots or displacement of the neighbouring teeth (Ericson and Kurol, 1988a, Ericson and Kurol, 2000, Falahat et al., 2008).

It has been suggested that if the primary ('baby' or 'milk') canine is extracted at an appropriate time in a child with a suspected palatally displaced canine, then the displaced tooth might spontaneously correct its position (Ericson and Kurol, 1988b) and the extraction of the baby canine when a clinician suspects that the adult canine is displaced has become accepted clinical practice (Short, 2009). This appears to be on the basis of one report of a series of 35 children who received the intervention and no control group (Ericson and Kurol, 1988b). Two recent systematic reviews have examined the evidence for the effectiveness of removal of the primary canine with the aim of correcting the eruption path of a palatally displaced canine. A recent systematic review published in The Cochrane Library in 2021 (Benson et al., 2021) noted that the evidence for any intervention to correct the eruption path of a displaced permanent canine is weak and further research is required. Numerous problems with the reported studies were identified by both reviews.

Other authors have suggested that using a RME (Rapid Maxillary expansion) or headgrear (EOT) to create sufficient space within the dental arch for the permanent canine tooth will encourage the tooth to erupt (Baccetti et al., 2011). This approach might be less traumatic to a child who may have had no experience of dental treatment, other than routine check-ups. If either or both approaches are shown to be effective then their widespread use would be advantageous to both the child and the healthcare provider, because the need for an operation, under general anaesthetic, to uncover the tooth and extensive brace treatment to straighten the tooth will be avoided.

DETAILED DESCRIPTION:
Design: A multicentre, parallel 3-group, randomised clinical trial. Setting: Orthodontic Departments in Sweden (5 centres), Germany (5 centres) and the UK (Sheffield).

Target Population: Children, aged 10-11 years. Inclusion criteria: One or both upper permanent canine teeth are not palpable or there is a pronounced difference in the eruption between the left and right side. Dental radiographs will be taken to confirm that the permanent tooth is displaced. Canines in sector 5 are going to be excluded from this trial.

Exclusion criteria: Buccal displacement of the canine(s), missing permanent lateral incisors; severe upper arch dental crowding (>2mm in each affected quadrant) or associated pathology.

Intervention: The trial will examine the effectiveness of early orthodontic intervention, either by removal of the baby canine tooth or opening space for the adult tooth, against no treatment.

Primary outcome • The proportion of young people who do not require surgery after 18 months from randomisation.

Secondary outcomes

* Cost effectiveness of the interventions
* Prevalence and severity of damage to surrounding teeth either due to the unerupted tooth or orthodontic intervention.

Sample size: A sample size calculation suggests that we will need to recruit 324 children (108 per group), assuming a dropout rate of 15%.

Research questions The study aim is to investigate whether early intervention, in children with one or both palatally displaced permanent maxillary canine, prevents the need for later more invasive, prolonged and costly surgical intervention.

Secondary research questions will include:

* What is the cost of early intervention compared with late intervention (surgery to uncover the tooth)?
* Is there a higher or lower incidence of damage to the surrounding teeth following early intervention?
* Are there any adverse effects of early intervention?

The trial efficacy objective will be to evaluate:

• The proportion of participants who have to undergo a surgical operation to uncover or expose the unerupted permanent canine after 18 months from randomisation (primary outcome).

Methods Population Children, aged 10-11 years with at least one palatally displaced maxillary permanent canine.

Interventions Participants will be randomised, using a centralised web-based system, with allocation stratified according to the position of the unerupted canine. The severity of displacement is important when deciding which treatment might be appropriate. Current practice is to extract the baby tooth in children with moderately displaced permanent teeth, but to retain the baby tooth if the permanent tooth is severely displaced. Canine teeth that are severely displaced towards the midline are thought to be less likely to respond to intervention than those nearer to the ideal position (Bazargani et al. 2014, Naoumova et al., 2015).

Young people with moderately displaced permanent canines (Sectors 2, 3 & 4 (Ericson and Kurol, 1988b), Figure below, will be allocated to one of 3 parallel arms:

* Control: no treatment;
* TrtA: open space between the lateral incisor and primary first molar/permanent premolar, to at least 9 mm, to ensure that there is sufficient space into which the canine can erupt; the space is to open whether with fixed appliance in the upper jaw and push coil or with RME
* TrtB: the primary canine(s) removed.

The allocation ratio within the stratum will be: Control: 1; TrtA: 1; TrtB:1. Data from previous studies suggest that in about 14% of young people with a palatally displaced canine the tooth is severely displaced towards the midline (Sectors 4, see ref above (Ericson and Kurol, 1988b)). For young people with a moderately displaced permanent canine there is some evidence that extracting the primary tooth might improve the position of the permanent tooth, hence the design of a three-arm trial. This will generate preliminary evidence of the relative efficacy between the two active arms. Patients with both upper canine teeth affected, but with different degrees of displacement, will be randomised according to the position of the most severely displaced tooth.

Comparator Those in the comparator group will have no treatment during the observation period of 18 months following diagnosis. Any necessary surgical or orthodontic treatment will be provided after this time if the permanent canine shows no signs of appearing in the mouth.

Outcomes The primary outcome will be the proportion of children who do not require surgery after 18 months from randomisation. This will be determined by the clinician treating the participants who will decide if the canine(s) is (are) in such a position that an orthodontic appliance can be placed without the need for surgical intervention. This will also be assessed, by independent judges, from masked clinical photographs taken at T2.

Secondary outcomes will include patient reported outcomes:

Incidence of Damage: Is there a higher or lower incidence of damage to the surrounding teeth following early intervention? Adverse Effects: Are there any adverse effects associated with early intervention?

* Quality of Life: How do children perceive their Oral Health-Related Quality of Life (OHrQoL) before, during and following early intervention, as assessed by the CPQ 11-14 and CHU9D?
* Cost-utility analysis: What is the cost of the different early interventions studied in relation to changes in HRQoL measured with CHU9D?

All outcomes are going to evaluated according to the intention-to-treat (ITT) analysis.

Proposed sample size and analyses The total number of patients required depends on the expected prevalence of the three strata. Assuming an effect size of 0.455 [ Nauomova et al., 2015] and further assuming a 15% drop-out, we will allocate 108 subjects to TrtA, 108 to TrtB and 108 to control (total 324), which gives a 80% power.

The primary outcome will be evaluated using a logistic regression with treatment (control vs TrtA or control vs TrtB) and strata as covariates. The same analysis will be used to evaluate the potential damage to surrounding teeth.

The economic analysis will be used to assess any differences in the cost effectiveness of early versus late intervention (surgical exposure). Costs of surgical exposures is going to be adapted from Björksved et al. [Björksved et al.; 2021].

Recruitment rate The recruitment rate per centre would be one participant every two months; therefore, to achieve a sample size of 300 participants in at least 15 centres would require 24 months.

Procedure Children with uni- or bilateral PDC:s meeting the inclusion criteria and their care givers/parents obtain information about the trial, both verbally and in writing. The children and their parents will be allowed at least one week to decide whether they wish to participate in the trial. After informed consent is obtained, the participants are randomly allocated to 1 of 3 groups. A computer-generated randomization is undertaken to ensure that there are equal numbers allocated to each group. Allocation concealment is held by one individual per centre, not involved with the trial.

In the TrtA group, the space creation will be achieved either through bonding fixed appliances in the upper jaw combined with the use of an open-coil or via RME (band on the first upper molars and arms stretching up to the first primary molars/ first premolars). The RME activation protocol is as follows: a single activation (0.25 mm) daily for a period of 14 days, followed by activation every other day until the point at which the palatal cusps of the maxillary first molars contacted the buccal cusps of the mandibular first molars).

Within Sweden, TrtB group is set to receive a space-maintaining appliance, a lingual arch, after the extraction of the primary canines. This is in order to preserve the arch perimeters throughout the observation period.

Study casts (preferably digital casts) at different timepoints (T0 = baseline, T1= 12 mon follow-up and T2 = 18 mon follow-up, see flowchart) are going to facilitate the monitoring of the space relationships in the dental arch.

Standardized panoramic radiographs at T0, T1 and T2 is going to be used to monitor the PDC:s angulation and potential improvement or worsening during the observations period of 18 months.

CBCT (cone beam computed tomography) at T0 and T2 are going to determine the presence or absence of root resorptions at baseline and T2 and the exact location of the PDC at baseline and at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* One or both upper permanent canine teeth are not palpable or there is a pronounced difference in the eruption between the left and right side. Dental radiographs will be taken to confirm that the permanent tooth is displaced. Canines in sector 5 are going to be excluded from this trial.

Exclusion Criteria:

* Buccal displacement of the canine(s), missing permanent lateral incisors; severe upper arch dental crowding (>2mm in each affected quadrant) or associated pathology.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 324 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Succeful eruption of the palatally displaced canines into the dental arch | 18 months after intervention
  The proportion of young people who do not require surgery after 18 months from randomisation.

SECONDARY OUTCOMES:
Cost effectiveness of the interventions | 18 months
  The proportion of young people who do not require surgery after 18 months from randomisation.
Prevalence and severity of damage to surrounding teeth either due to the unerupted tooth or orthodontic intervention. | 18 months
  Prevalence of root resorptions to the adjacent teeth measured with computed tomography
Oral Health related Quality of Life | At baseline, 6 months and 18 months
  Using Child Perception Questionnaire
Cost-utility analysis | At baseline, 6 months and 18 monts
  Using Child Health Utility 9D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Bazargani, DDS, PhD, Principal Investigator — Gothenburg University, Gothenburg, Sweden
Locations (3):
- Private practice, Traben-Trarbach, Germany
- Gothenbrug University, Gothenburg, Sweden
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No